CLINICAL TRIAL: NCT07025252
Title: Outcomes for VersaWrap in Achilles Tendon Repair
Status: Enrolling by invitation | Type: Observational
Sponsor: Research Source (Network)
Responsible Party: Sponsor
Other Study IDs: TP-068
Record Dates: First submitted 2025-06-09; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Achilles Tendon Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- VersaWrap: All enrolled patients will received VersaWrap applied prior to surgical closure on the affected tendon.
  Interventions: Device: VersaWrap

INTERVENTIONS:
Device: VersaWrap — VersaWrap is applied to the affected tendon to allow post-operative gliding.

SUMMARY:
The purpose of this study is to evaluate the efficacy on the use of VersaWrap® in surgery of the foot and ankle. VersaWrap is designed to allow tendon gliding and to protect tendon gliding postoperatively

DETAILED DESCRIPTION:
This is a prospective, multi-center, controlled case series evaluating the use of VersaWrap in surgeries of the foot and ankle. Patients identified by the Investigator in his practice as needing surgery for an Achilles primary or elective insertional repair and meeting all the inclusion and none of the exclusion. Patients will consent to participating in the study, prior to any study procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Patients that require surgery for Achilles primary or elective insertional repair. Note: primary repair must be conducted within 6 weeks of injury. Additional repairs may be conducted during surgery, confirm with study Sponsor prior to enrollment. Insertional repairs due to trauma are not eligible.
2. Able to understand the requirements of the study, provide a written consent, and willing to comply with the study protocol
3. Age ≥18 years and <90 years at the time of surgery

Exclusion Criteria:

1. Investigator determines that the subject is unlikely to comply with the requirements of the study
2. Active systemic infection or infection at the location planned surgery
3. Uncontrolled diabetes
4. Prior Achilles surgery on either ankle
5. Active or suspected malignancy. If symptom free for 2 years, patients with prior malignancy may be included
6. Morbid obesity defined as a body mass index > 40
7. Pregnant or have plans to become pregnant in the next year
8. Currently a prisoner
9. Autoimmune disorders that impact the musculoskeletal system (e.g., lupus, rheumatoid arthritis; ankylosing spondylitis)
10. Medications that could interfere with fusion or other bone/soft tissue healing (e.g., anticipated continued use of systemic steroid medication postoperatively)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who meet the following inclusion criteria and none of the exclusion criteria will be enrolled in the study. A patient is considered enrolled upon placement of the VersaWrap during the surgical procedure. If the surgeon decides intra-operatively not to utilize the VersaWrap, the patient will be considered a screen failure.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Skin Excursion | 12 months post surgery
  Skin excursion will be measured by examining the movement that is regularly repeated in a portion of involved skin in comparison to movement of the skin in the peroneal region of the contralateral foot. A ruler will be utilized to measure the up and down movement at the center of the skin excision, to determine the exact amount of excursion of the center of the wound.
Range of Motion (ROM) | 12 months post surgery
  Standing dorsi- and plantarflexion of the affected and contralateral ankle will be measured using a handheld goniometer, referencing the long axis of the fibula and fifth metatarsal shaft. Both passive and active range of motion will be captured. The greater the ROM the better the outcome.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - UC Davis Foot and Ankle Orthopaedics Clinic, Sacramento, California
  - Rothman Orthopaedics Institute, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No